CLINICAL TRIAL: NCT02663817
Title: DMH-Based Plan Evaluation and Inverse Optimization in Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ivaylo Mihaylov, PhD, DABR, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20130751; R01CA163370 (NIH)
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Cancer; Lung Cancer; Prostate Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Prostatic Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- IMRT (Experimental): Study participants being treated according to the standard of care with intensity modulated radiotherapy (IMRT). Several CT scans will be performed for each enrolled subject: one before the radiotherapy course for patient treatment planning purposes (as part of the standard of care), one during the radiotherapy treatment course (between fraction 10 and 20), and one at follow up visit or at least 6 weeks post-radiotherapy treatment (whichever comes first).
  Interventions: Device: CT Scan

INTERVENTIONS:
Device: CT Scan
  Other Names: Computed Tomography Imaging Scan

SUMMARY:
The hypotheses of the study are as follows:

* Mass-based inverse optimization in radiotherapy treatment planning will result in a reduction of normal tissue and organs at risk (OAR) doses for desired prescription therapeutic doses to the targets.
* Dose-mass histograms (DMHs) may be more relevant to radiotherapy treatment planning and treatment plan assessment than the standard of care, realized through dose-volume histograms (DVHs)

DETAILED DESCRIPTION:
Cancer patients continue to represent a challenging disease population, which faces rather poor prognosis with current treatment planning and delivery practices. Venues for a potential dose escalation and/or increased healthy tissue sparing, through innovative therapeutic approaches for those patients, are clearly needed. Current state of the art radiotherapy treatment planning relies on the dose-volume-histogram (DVH) paradigm, where doses to fractional (most often) or absolute volumes of anatomical structures are employed in both optimization and plan evaluation process. It has been argued however, that the effects of delivered dose seem to be more closely related to healthy tissue toxicity (and thereby to clinical outcomes) when dose-mass-histograms (DMHs) are considered in treatment plan evaluation.

The investigators propose the incorporation of mass and density information explicitly into the cost functions of the inverse optimization process, thereby shifting from DVH to DMH treatment planning paradigm. This novel DMH-based intensity modulated radiotherapy (IMRT) optimization aims in minimization of radiation doses to a certain mass, rather than a volume, of healthy tissue. The investigators' working hypothesis is that DMH- optimization will reduce doses to healthy tissue substantially. In certain cases, with extensive, difficult to treat disease, lower doses to healthy tissue can be used for isotoxic dose escalation, which may result in an increase in estimated loco-regional tumor control probability.

To test the study hypothesis, the investigators will pursue the following specific aims:

* (1) Develop the theoretical and computational framework of the DMH-based IMRT optimization. This framework will incorporate 3D and 4D IMRT as well as 3D volumetric modulated arc (VMAT) planning for different anatomical sites.
* (2) Investigate different parametric forms for DMH-optimization functions. The ultimate goal would be the simultaneous minimization of healthy tissue doses and/or escalation of therapeutic doses, without violating the established dosimetric tolerances for healthy anatomical structures.
* (3) Practical implementation and application of this novel optimization paradigm, where virtual clinical trials for cohorts of lung, head-and-neck, and prostate cancer cases will be performed.

Statistical significance of the DMH-optimization dosimetric improvements over standard of care DVH-optimization will be quantified. Prospective 3D and 4D CT data collection will be used to study the interactions between tumor time-trending changes and DMH-based optimization results. 4D CT data will also be used to investigate and quantify the correlation between DMH-based end points and the loss of pulmonary function during and after radiotherapy treatment. The deliverability (with the existing radiotherapy treatment equipment) of the investigators' 3D VMAT and 3D/4D IMRT plans will be experimentally verified, thereby paving the road for initiation of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed head-and-neck, lung, or prostate tumors.
* Patients who will be treated with radiation therapy or concurrent chemoradiation therapy.
* Gross Tumor Volume (GTV) or resection cavity must be visible on CT such that it can be delineated as a target for radiotherapy.
* Patients who are able to understand the investigational nature of this study and agree to sign a written informed consent document.

Exclusion Criteria:

* Pregnant or nursing women will not participate. Women of reproductive potential must be offered a pre-treatment pregnancy test and informed of the need to practice an effective contraceptive method during the therapy.
* Patients younger than 18 years.
* Patients whose size and weight would not allow CT scanning.
* No vulnerable populations (fetuses, pregnant women, children, prisoners) will be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivaylo Mihaylov, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMRT
Started | 52
Completed | 50
Not Completed | 2
Not completed — Screen failure | 2

BASELINE CHARACTERISTICS:
Arm/Group | IMRT
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 39
  More than one race | 2
  Unknown or Not Reported | 2
Disease site [Count of Participants; unit: Participants]
  Head and neck | 27
  Prostate | 9
  Lung | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Radiation Dose to Healthy Human Tissue.
Description: The study is computational in nature. A new treatment planning paradigm is proposed, where from the newly proposed treatment plans, and the treatment plans generated with the standard of care, radiation doses to different organs and tissues would be derived. Radiotherapy toxicity (to healthy human tissue) is proportional to radiation dose - more radiation dose results in higher toxicity. Thereby, if radiation dose is decreased, the toxicity would also be decreased. The dosimetric differences which the investigators observe between the standard of care and their novel optimization approach are reported as percent change with respect to the standard of care.
Time Frame: Baseline, up to three years.
Population: Two participants with prostate cancer were screen failures.
Measure: Mean (Full Range); unit: Percent change in radiation dose
Groups:
- IMRT Lung: Study participants being treated according to the standard of care with intensity modulated radiotherapy (IMRT) for Lung cancer.
- IMRT Prostate: Study participants being treated according to the standard of care with intensity modulated radiotherapy (IMRT) for Prostate cancer.
- IMRT Head and Neck: Study participants being treated according to the standard of care with intensity modulated radiotherapy (IMRT) for Head-and-Neck cancer.
Arm/Group | IMRT Lung | IMRT Prostate | IMRT Head and Neck
Number analyzed (Participants) | 16 | 7 | 27
Percent change in radiation dose
  Dmh - Heart: number analyzed (Participants) | 16 | 0 | 0
  Dmh - Heart | 3.0 [-4.9 to 8.0] |  |
  Dmh - Spinal Cord: number analyzed (Participants) | 16 | 0 | 0
  Dmh - Spinal Cord | 31.0 [-8.0 to 67.0] |  |
  Dmh - Esophagus: number analyzed (Participants) | 16 | 0 | 0
  Dmh - Esophagus | 25.0 [-2.6 to 61.0] |  |
  Dmh - Lungs: number analyzed (Participants) | 16 | 0 | 0
  Dmh - Lungs | 2.0 [-3.0 to 6.0] |  |
  Energy - Heart: number analyzed (Participants) | 16 | 0 | 0
  Energy - Heart | 11.0 [0.1 to 44.7] |  |
  Energy - Spinal Cord: number analyzed (Participants) | 16 | 0 | 27
  Energy - Spinal Cord | 24.0 [-8.0 to 63.0] |  | 7.0 [-5.0 to 27.0]
  Energy - Esophagus: number analyzed (Participants) | 16 | 0 | 0
  Energy - Esophagus | 16.0 [-2.6 to 39.7] |  |
  Energy - Lungs: number analyzed (Participants) | 16 | 0 | 0
  Energy - Lungs | 10.0 [-3.0 to 21.0] |  |
  Energy for HN - Brainstem: number analyzed (Participants) | 0 | 0 | 27
  Energy for HN - Brainstem |  |  | 11.0 [-5.0 to 34.1]
  Energy for HN - Larynx: number analyzed (Participants) | 0 | 0 | 27
  Energy for HN - Larynx |  |  | 9.0 [-7.0 to 21.0]
  Energy for HN - Lt Parotid: number analyzed (Participants) | 0 | 0 | 27
  Energy for HN - Lt Parotid |  |  | 14.0 [-17.0 to 38.0]
  Energy for HN - Rt Parotid: number analyzed (Participants) | 0 | 0 | 27
  Energy for HN - Rt Parotid |  |  | 13.0 [-7.0 to 38.5]
  Energy Prostate - Bladder D15: number analyzed (Participants) | 0 | 7 | 0
  Energy Prostate - Bladder D15 |  | 2.0 [-2.6 to 10.6] |
  Energy Prostate - Bladder D25: number analyzed (Participants) | 0 | 7 | 0
  Energy Prostate - Bladder D25 |  | 6.5 [-5.5 to 30.0] |
  Energy Prostate - Rectum D15: number analyzed (Participants) | 0 | 7 | 0
  Energy Prostate - Rectum D15 |  | 1.7 [-6.0 to 9.7] |
  Energy Prostate - Rectum D25: number analyzed (Participants) | 0 | 7 | 0
  Energy Prostate - Rectum D25 |  | 5.0 [-1.2 to 11.5] |
  Energy Prostate - Rt Femur D10: number analyzed (Participants) | 0 | 7 | 0
  Energy Prostate - Rt Femur D10 |  | 32.5 [-0.8 to 71.0] |
  Energy Prostate - Lt Femur D10: number analyzed (Participants) | 0 | 7 | 0
  Energy Prostate - Lt Femur D10 |  | 32.7 [-0.6 to 78.0] |

ADVERSE EVENTS:
Description: No adverse events were collected in this protocol
Arm/Group | IMRT
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT02663817/Prot_SAP_000.pdf